CLINICAL TRIAL: NCT00318487
Title: Bilateral Sinus Floor Augmentation in Conjunction With Immediate Implant Loading - A Clinical and Histomorphometric Follow-Up Study on 3i Dental Implants
Brief Title: Bilateral Sinus Floor Augmentation in Conjunction With Immediate Implant Loading - Study on 3i Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/126
Record Dates: First submitted 2006-04-11; First posted 2006-04-26 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Mouth, Edentulous
Keywords: Dental implants
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bilateral sinus augmentation (Experimental)
  Interventions: Procedure: Bilateral sinus augmentation with immediately loaded dental implants

INTERVENTIONS:
Procedure: Bilateral sinus augmentation with immediately loaded dental implants — Bilateral sinus augmentation with immediately loaded dental implants will be used.

SUMMARY:
Fifteen (15) patients completely edentulous in the maxilla will be treated with 8 dental implants. The total treatment will be done in 2 stages to allow, within the same group, a study of two different approaches. Miniscrews that can be functionally loaded will be provided by 3i with the design and surface textures as wanted by the study sponsor.

DETAILED DESCRIPTION:
The department of oral surgery in Ghent has a lot of patients for bilateral sinus lift procedures. The group of patients should have enough bone for installation of 4 dental implants in the area 14-24. In this region 4 implants will be installed and immediate loading with a provisional acrylic (metal reinforced) bridge will be provided. The survival and success of the implants immediate functional loading will be studied (interest point 1). Two different implant surfaces are used in the study to be compared (interest point 2) in relation to peri-implant parameters, radiographical healing, and success criteria at the same time bilateral sinus lifting is performed. One sinus is filled with a mixture of iliac crest bone and Bio-Oss (Geistlich Germany), and the second sinus is filled with calvarial skull bone and Bio-oss. The latter bone combination is appreciated clinically by the surgeons since it leads to a subjectively better implant stability. This, however, remains to be investigated. This study can compare both harvesting techniques and evaluate clinical treatment outcome (interest point 3). Normally, there is a certain waiting time after sinus lifting before dental implants are installed. Recently, however, some literature abstracts indicate that immediate placement of the implants in the sinus lifted bone can be successful. However, this is not done with immediate functional loading. We propose to install in total 6 miniscrews, 2 in each sinus lift area. Four will be loaded immediately and connected rigidly to the other 4 normal sized implants. Actually the immediate loaded bridge will be supported, in total, by 4 normal and 4 miniscrew implants. Four months after loading, the 4 loaded miniscrews are removed with a trephine drill in order to examine soft-tissue healing, bone-implant contact, and bone healing by means of histomorphometry. Since the implants are in cortical bone + sinus lifted bone, it will be possible to examine the given implant surface under immediate loading in both bone conditions (interest point 4). Immediately after removing the miniscrews, they are replaced by the normal sized implants. One side will be randomly assigned for immediate non-functional loading, the other side will be assigned to a non-loaded condition. With this latter design we can mimic the partial sinus lift condition as it is often done 4 months after sinus lifting - the classical procedure. At the time of exposing the implants of the 2-stage procedure, the miniscrews are removed. This gives us an idea of bone healing of an implant installed 4 months after sinus lifting and kept additionally unloaded for 4 months. This gives us histology of immediately loaded implants in healed sinus lifted bone (interest point 5).

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with a full removable denture in the maxilla.
* Subjects must have enough bone to install 4 dental implants in region 14 to 24 and are in need of a sinus lifting procedure in the posterior mandible (region 18-15 + 25-28).

Exclusion Criteria:

* Patients with compromised healing capacities such as cancer patients and diabetes patients.
* Smokers are excluded when smoking > 12 cigarettes per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-09-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of 3i dental implants installed simultaneously with a sinus lift procedure and immediately loaded | 4 months
Comparison of sinus lift with autogenous iliac crest bone + Bio-Oss and sinus lift with an autogenous calvarial skull bone + Bio-Oss | 4 months
Installation of implants Prevail and Certain in sinus lift area and naturally healed (non-lifted) bone | 4 months
Histological comparison between immediately loaded implants in sinus lifted bone versus normal bone | 4 months
Histological comparison at various time intervals | 4 months
Histologic findings: integration of the graft, amount of new bone formation, survival and success of the implant, and osseointegration of implant | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be